CLINICAL TRIAL: NCT03349125
Title: Effects of Cervical Bracing on Elderly Patients With Dysphagia
Brief Title: Study: C-Collar and Dysphagia
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-0222; A539772 (Other: UW Madison); SMPH/SURGERY/SURGERY*SP (Other: UW Madison)
Record Dates: First submitted 2017-10-25; First posted 2017-11-21 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Dysphagia
Keywords: Cervical Brace; Elderly; Dysphagia; VFSS; Videoflouroscopy; Swallow Problems
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Collar On: Individuals who have been referred for videoflouroscopic swallow study (VFSS) as per standard of care, with a stable cervical injury, will have trials of liquids and solids with the Cervical Brace (Collar) on.
  Interventions: Behavioral: Collar On
- Collar Off: Individuals who have been referred for videoflouroscopic swallow study (VFSS) as per standard of care, with a stable cervical injury, will have trials of liquids and solids with the Cervical Brace (Collar) off.
  Interventions: Behavioral: Collar Off

INTERVENTIONS:
Behavioral: Collar On
  Groups: Collar On
Behavioral: Collar Off
  Groups: Collar Off

SUMMARY:
The purpose of this study is to characterize oral-pharyngeal swallow function with the guidance of videofluoroscopy under two conditions, with and without cervical bracing, in patients determined to have dysphagia.

DETAILED DESCRIPTION:
According to the National Cervical Spinal Cord Injury Statistical Center, 12,000 patients experience acute spinal cord injury (SCI) in the United States annually. It is reported that 16% to 55% of patients with a cervical spinal cord injury (SCI) present with dysphagia which compromises their ability to eat and drink safely as well as their quality of life. Based on previous research, Dysphagia can also result in respiratory complications, particularly pneumonia, which is the most common cause of death in cervical SCI patients. The contribution of swallowing impairment, and associated aspiration risks, to respiratory illnesses and mortality in patients with SCI are unknown. As a first step, the investigators will identify the nature (type of swallowing impairment such as swallow delay, pharyngeal residue, penetration or aspiration) and frequency of occurrence of swallowing impairments in elderly patients with injury to the cervical spinal region. Further, the investigators will determine the effects of standard medical care, specifically, surgical bracing, on swallow function in patients post-cervical SCI.

Patients with SCI present with a range of impairments in the oral and pharyngeal phases of the swallow. These result both from the effects of trauma and medical/surgical management of injury on anatomy and physiology of the swallow mechanism. Earlier studies postulate that Acute SCI can result in reduced base of tongue movement, delayed pharyngeal swallow response, decreased hyolaryngeal excursion with subsequent decrease in cricopharyngeal opening, and pharyngeal wall dysfunction. These swallowing impairments are particularly devastating in older patients who lack the functional reserve to overcome these neuroanatomical insults. Consequently, there is an increased prevalence of dysphagia in the elderly patients with SCI.

Medical and surgical management of SCI can also negatively impact swallow function. Many patients will require neck immobilization following injury. Neck extension, chin or head retraction secondary to cervical bracing may increase the risk or severity of dysphagia by changing the mechanics of swallowing. In addition, fixation at a ninety-degree angle limits the natural flexion or range of movement a patient employs during deglutition. Studies have found that cervical orthoses impacts swallowing physiology in healthy adults. An earlier study reported changes in point of initiation of the swallow, laryngeal penetration, pharyngeal residue and hyoid bone movement. One would expect changes to be more significant in patients with dysphagia, and likely more remarkable in the elderly population who unfortunately, have the highest incidence of cervical SCI. Given the risk factors for dysphagia and pulmonary complications in this population, it is imperative that thorough evaluation of oral-pharyngeal swallow function be completed. However, there is little research addressing the impact of cervical bracing on patients with dysphagia at any age. The study team here aims to determine if cervical bracing contributes to severity of dysphagia.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatients receiving treatment for a spine injury
2. Treating physician's approval that cervical cervical spinal column injury is stable
3. Approval for collar removal by treating physician during VFSS
4. Adults 60 and over.
5. All races.
6. Males and females.
7. Glasgow coma scale of 13 or greater.

Exclusion Criteria:

1. History of oral-pharyngeal dysphagia.
2. Neurologic disorders associated with dysphagia including dementia, Parkinson's disease, multiple sclerosis, stroke, and ALS.
3. Pharyngeal/laryngeal surgery or head/neck radiation treatment.
4. Glasgow coma scale of less than 13 at time of evaluation.
5. Patient's with a tracheotomy.
6. Barium intolerance.
7. Patients who lack the capacity to consent on their own behalf

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients with dysphagia in a cervical brace.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2013-09-17 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2018-04-05 (Actual)

PRIMARY OUTCOMES:
To identify aspiration between study conditions (with and without a collar). | Comparing aspiration presence between two study conditions (with and without a cervical collar). Data will be reported at the end of study completion, an average of 1 year.
  Measures of dysphagia aspiration (Y/N) and will be obtained in subjects both with and without a collar during the swallow evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Jodi Hernandez, MS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States